CLINICAL TRIAL: NCT04600830
Title: Evaluation of the Effectiveness of Dry Needling Against Foam Roller in the Short Term, Healthy Athletes With Reduced Mobility of the Ankle Joint
Brief Title: Evaluation of the Effectiveness of Dry Needling Versus Foam Roller
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2019 - 2020/062
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Myofascial Pain Syndromes; Dry Needling
Keywords: Dry needling; Myofascial pain syndromes; Ankle joint
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A simple blind masking will be carried out to reduce biases in the interpretation of the results. The researchers responsible for the observation, measurement of the ankle ROM and Counter Movement Jump, will not be informed of the treatment performed at the time of immediate post-treatment and post-treatment at 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental): Dry needling will be applied to the myofascial trigger points of the gastrocnemius muscle. With the dry needle (0.3 x 40 mm. Myofib, Toledo, Spain). Thus, insert the needle until you get the first twitch response. Once the first twitch response is obtained, the needle will move about 2-3 mm vertically quickly. Twenty-five insertions without leaving the skin. The approximate frequency of 1 Hz for 25 to 30 seconds.
  Interventions: Procedure: Dry needling
- Foam Roller Group (Active Comparator): The myofascial self-release technique with the FR Black Roll PRO (Bottighogen, Switzerland). The subject will move his body in the same direction as the muscle fibers, using his hands to propel and get the roller to slide back and forth. The device will only be applied at the muscular level, avoid the area of the Achilles tendon. It will be repeated on the contralateral leg. A total of three 60-second steps is executed on each leg and a 30-second break between both.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Intervention with deep dry needling on latent myofascial trigger points (MTrPs) in gastrocnemius muscle.

SUMMARY:
To compare the effects of dry needling and Foam roller in myofascial trigger points. Needling has been shown to decrease pain in the short term; however, its effects on muscle force production are unclear. There are differences between dry needling and foam roller after treatment?

DETAILED DESCRIPTION:
Background: It has been shown that the decrease of the range of motion in the ankle, due to the presence of latent trigger points in the gastro-sole complex, can affect performance, as well as being a predisposing factor to injury. Objective: To compare the effects of Dry Needling and Foam roller in healthy athletes with limited dorsal ankle flexion by the presence of latent trigger points. Material and methods: This is a clinical trial, single-blind experimental study. The sample will have a total of 44 students, volunteers, healthy of the degree of physiotherapy of the the investigator's university (UCV). Participants who meet the inclusion criteria will be randomly assigned in two groups: Group 1 or Dry Needling (N = 22) and Group 2 or Foam Roller (N = 22). The range of motion of ankle will be assessed through the Leg Motion system (Check Your Motion®, Albacete, Spain). Assessed thought Ankle Test (post-intervention and 24 hours later). The reference values to consider the decreased ankle ROM will be <11.5 cm, <35º measured with Easy Angle® digital goniometer (Meloq AB, Sweden) and/or if it has a difference of 1.5 cm between both extremities. Thus, the effect on previous activity performance will be assessed thought the Counter Movement Jump. Data analysis: Once the distribution of the sample is determined, a descriptive analysis of the data will be carried out and an ANOVA of repeated measures. Will be used to compare the data found in the two groups that make up the study taking into account a 95% CI and an error less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Students of physiotherapy degree of the university
* All participants who present restriction on active ankle dorsiflexion (<35º).
* They must be diagnosed through manual therapy of latent PG in the gastro-soleus complex.

Exclusion Criteria:

* Subjects suffering from belonephobia
* Pathology of connective tissue
* Coagulation problems
* Lymphatic disorders
* Diabetes
* Surgical history in the lower limb (last 12 months)
* Prior treatment with dry needling (last 6 months)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) | 48 hours
  Range of motion (ROM) is a key measurement to help in detecting and diagnosing musculoskeletal deficits, monitoring treatment progression, and guiding the treatment plan. Measurement of ROM is a relevant point and an important item of the joint evaluation process when using any ankle scoring system as part of the ankle and ankle joint evaluation. ROM of ankle joint in load PRE, POST treatment and POST 24 hours after of intervention.

SECONDARY OUTCOMES:
Lunge / Ankle Test Test | 48 hours
  he Weight-bearing lunge test (WBLT) or Dorsiflexion Lunge Test (DFT) is used to assess the dorsiflexion range of movement (DROM) at the ankle joint. Participants are instructed to lunge forward until their knee touches the wall (vertical line). The heel is required to remain in contact with the floor at all times. The foot is moved away from the wall to the point where the knee can only make slight contact with the Wall.
Counter Movement Jump (CMJ) | 48 hours
  The countermovement jump (CMJ) is a simple, practical, valid, and very reliable measure of lower-body power. This suggests that performances in the CMJ are linked with maximal speed, maximal strength, and explosive-strength. When the CMJ is performed using the arm-swing, performances can be ≥10% higher than when they include no arm-swing. Contact mats, force platforms, accelerometers, high-speed cameras, and infrared platforms have all been shown to provide a valid and reliable measure of CMJ performance - though force platforms are considered as the 'gold-standard'.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Vicente, Principal Investigator — Fundacion UCV
Locations (1):
- Juan Vicente Mampel, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grieve R, Clark J, Pearson E, Bullock S, Boyer C, Jarrett A. The immediate effect of soleus trigger point pressure release on restricted ankle joint dorsiflexion: A pilot randomised controlled trial. J Bodyw Mov Ther. 2011 Jan;15(1):42-9. doi: 10.1016/j.jbmt.2010.02.005. Epub 2010 Mar 23. PMID 21147417
- [Background] Gerwin RD. A review of myofascial pain and fibromyalgia--factors that promote their persistence. Acupunct Med. 2005 Sep;23(3):121-34. doi: 10.1136/aim.23.3.121. PMID 16259310
- [Background] de Benito AM, Valldecabres R, Ceca D, Richards J, Barrachina Igual J, Pablos A. Effect of vibration vs non-vibration foam rolling techniques on flexibility, dynamic balance and perceived joint stability after fatigue. PeerJ. 2019 Nov 26;7:e8000. doi: 10.7717/peerj.8000. eCollection 2019. PMID 31788353
- [Background] Calatayud J, Martin F, Gargallo P, Garcia-Redondo J, Colado JC, Marin PJ. The validity and reliability of a new instrumented device for measuring ankle dorsiflexion range of motion. Int J Sports Phys Ther. 2015 Apr;10(2):197-202. PMID 25883868
- [Background] Grieve R, Goodwin F, Alfaki M, Bourton AJ, Jeffries C, Scott H. The immediate effect of bilateral self myofascial release on the plantar surface of the feet on hamstring and lumbar spine flexibility: A pilot randomised controlled trial. J Bodyw Mov Ther. 2015 Jul;19(3):544-52. doi: 10.1016/j.jbmt.2014.12.004. Epub 2014 Dec 18. PMID 26118527